CLINICAL TRIAL: NCT05477524
Title: A Phase 3, Multicenter, Placebo-Controlled, Randomized, Observer-Blinded Trial to Evaluate the Efficacy, Safety, Tolerability, Immunogenicity, and Lot Consistency of a 6-Valent OspA-Based Lyme Disease Vaccine in Healthy Participants ≥5 Years of Age
Brief Title: An Efficacy, Safety, Tolerability, Immunogenicity, and Lot-Consistency Clinical Trial of a 6-Valent OspA-Based Lyme Disease Vaccine (VLA15)
Acronym: VALOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4601003; 2023-509105-72-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-07-05; First posted 2022-07-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Lyme Disease
Keywords: VLA15; Lyme Borreliosis; Vaccine; Tick
MeSH Terms: conditions — Lyme Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VLA15 Lot 1 (3-dose primary vaccination series and booster dose) (Experimental): Shot in the deltoid muscle (preferable in the nondominant arm)
  Interventions: Biological: VLA15
- VLA15 Lot 2 (3-dose primary vaccination series and booster dose) (Experimental): Shot in the deltoid muscle (preferable in the nondominant arm)
  Interventions: Biological: VLA15
- VLA15 Lot 3 (3-dose primary vaccination series and booster dose) (Experimental): Shot in the deltoid muscle (preferable in the nondominant arm)
  Interventions: Biological: VLA15
- Placebo (3-dose primary vaccination series and booster dose) (Placebo Comparator): Shot in the deltoid muscle (preferable in the nondominant arm)
  Interventions: Other: Saline

INTERVENTIONS:
Biological: VLA15 — Shot in the deltoid muscle (preferable in the nondominant arm)
  Arms: VLA15 Lot 1 (3-dose primary vaccination series and booster dose); VLA15 Lot 2 (3-dose primary vaccination series and booster dose); VLA15 Lot 3 (3-dose primary vaccination series and booster dose)
Other: Saline — Shot in the deltoid muscle (preferable in the nondominant arm)
  Arms: Placebo (3-dose primary vaccination series and booster dose)

SUMMARY:
The main purpose of this clinical study is to evaluate a 6-valent OspA-based Lyme disease vaccine (VLA15) for prevention of Lyme disease within North America and Europe. Approximately 9,400 healthy participants (this number excludes participants from 8 sites which were terminated for quality issues) 5 years and older will be recruited from areas with high levels of endemic Lyme disease to receive VLA15 or placebo (an inactive substance consisting of saltwater). Each participant will have about a 50% chance of receiving VLA15 and about a 50% chance of receiving placebo. A subset of participants will receive VLA15 from 3 different lots or placebo (1:1:1:3 ratio) to assess lot equivalence.

Participants will receive a 3-dose primary vaccination series at about 0, 2, and 5 to 9 months and then receive a booster dose about 12 months after end of primary vaccination series. Vaccination of participants will occur at a time of year such that the primary series is completed before the peak Lyme disease season followed by a booster dose just prior to the beginning of the second Lyme disease season. A subset of participants will be followed for a third Lyme disease season.

Comparison will be made between the Lyme disease cases of people receiving the study vaccine to those of the people who are not. This will help us determine if the study vaccine is safe and effective.

If enrolled, participants will need to visit the research site at least 7 times during the study, and for a subset of participants up to 9 times. There will also be at least 5 telephone contacts. It is expected that each participant will take part in this study for up to about 2 and a half years. The subset of participants followed for a third Lyme disease season will take part in this study for up to about to 3 and a half years.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who reside in areas with endemic Lyme disease and who lead lifestyles that put them at increased risk for Lyme disease. For example, this could include, but not be limited to:
* Individuals who work in B burgdorferi-infected/tick-infested areas, especially those with occupations that may be associated with higher risk of exposure, such as landscaping, forestry, and wildlife and parks management.
* Individuals who pursue recreational activities such as hiking, camping, fishing, hunting, jogging, or gardening in such areas.
* Individuals who live on land plots with tree lines and come into contact with these trees regularly.
* Individuals who have dogs that regularly are outdoors and frequently return with attached ticks.
* Individuals who participate in activities in areas with tall grass, smaller wooded areas beside forests, open fields, lakesides, and riversides.

Key Exclusion Criteria:

* Any female participants that are pregnant (or have a positive urine pregnancy test) or are breastfeeding.
* Any diagnosis of Lyme disease within the past 3 months.
* Any history of Lyme carditis, neuroborreliosis, or arthritis, or other disseminated Lyme disease regardless of when diagnosed.
* Known tick bite within the past 4 weeks.
* Newly developed or unstable underlying conditions that may interfere with the assessment of Lyme disease, including but not limited to chronic arthralgia/arthritis, second/third-degree AV heart block, chronic pain syndromes, and chronic skin conditions that reduce the ability to detect cutaneous manifestations of Lyme disease.
* Any unstable autoimmune condition with a manifestation (eg, arthritic and neurologic) that may interfere with the assessment of Lyme disease.
* Chronic systemic doxycycline or minocycline or other tetracycline class drug use for acne or any other chronic suppressive antibiotics used to treat other conditions.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12547 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-12-26 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Relative incidence rate reduction of confirmed Lyme disease cases in the VLA15 group compared to the placebo group | Beginning 1 month after receiving the booster dose (28 days after receiving the booster dose through the end of the Lyme disease season following the booster dose (end of October)).
  A confirmed case of Lyme disease, caused by B burgdorferi sensu lato, is defined as a clinically suspected case of Lyme disease that is confirmed by PCR, culture, microbial cell-free B burgdorferi-specific DNA sequencing, or serological antiborrelial antibody assay, and finally assessed and confirmed to be a case by the independent Adjudication Committee
Percentage of participants reporting local reactions | Within 7 days following each study intervention administration
Percentage of participants reporting systemic events | Within 7 days following each study intervention administration
Percentage of participants reporting adverse events (AEs) | Through 1 month following each study intervention administration
Percentage of participants reporting newly diagnosed chronic medical conditions (NDCMCs) | Through study completion, up to approximately 42 months.
Percentage of participants reporting serious adverse events (SAEs) | Through study completion, up to approximately 42 months.
Geometric mean ratio (GMR) of anti-OspA titers for each serotype (ST1-ST6) for Lot 1 to Lot 2 | At 1 month after completion of the primary series and the booster dose
Geometric mean ratio (GMR) of anti-OspA titers for each serotype (ST1-ST6) for Lot 1 to Lot 3 | At 1 month after completion of the primary series and the booster dose
Geometric mean ratio (GMR) of anti-OspA titers for each serotype (ST1-ST6) for Lot 2 to Lot 3 | At 1 month after completion of the primary series and the booster dose
Geometric mean ratio (GMR) of anti-OspA titers for each serotype (ST1-ST6) | At 1 month after completion of the booster dose
  Immunobridging objective to determine non-inferiority between 5-17 year old and 18-44 year old participant strata.

SECONDARY OUTCOMES:
Vaccine efficacy among participants enrolled from North American sites | Through the end of the Lyme disease season beginning 1 month after receiving the booster dose (28 days after completion of the booster dose until end of October)
  A confirmed case of Lyme disease, caused by B burgdorferi sensu lato, is defined as a clinically suspected case of Lyme disease that is confirmed by PCR, culture, microbial cell-free B burgdorferi-specific DNA sequencing, or serological antiborrelial antibody assay, and finally assessed and confirmed to be a case by the independent Adjudication Committee
Vaccine efficacy among participants after primary series | Through the end of the Lyme disease season beginning 1 month after completing the primary series (28 days after completion of the primary series until end of October)
  A confirmed case of Lyme disease, caused by B burgdorferi sensu lato, is defined as a clinically suspected case of Lyme disease that is confirmed by PCR, culture, microbial cell-free B burgdorferi-specific DNA sequencing, or serological antiborrelial antibody assay, and finally assessed and confirmed to be a case by the independent Adjudication Committee

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (119):
- United States (73):
  - Care Access - Essex, Essex, Connecticut
  - Care Access Mobile Site, New London, Connecticut
  - Stamford Health Medical Group, Stamford, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Care Access - Farmington, Farmington, Maine
  - Pen Bay Medical Center, Rockport, Maine
  - Johns Hopkins, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Rockland Physician Practice and Research Group, Lutherville, Maryland
  - Sumit Bhutani MD LLC, Westminster, Maryland
  - Woodholme Gastroenterology Associates, Westminster, Maryland
  - Pediatric Associates of Fall River, Fall River, Massachusetts
  - Care Access - Lakeville, Lakeville, Massachusetts
  - Care Access - Melrose, Melrose, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Care Access - Briarpatch and Mobile Site, Nantucket, Massachusetts
  - Care Access - Nantucket, Nantucket, Massachusetts
  - Care Access Mobile Site, Nantucket, Massachusetts
  - South Shore Medical Center, Norwell, Massachusetts
  - Care Access - Hingham, Rockland, Massachusetts
  - Sisu BHR, Springfield, Massachusetts
  - Care Access - Wareham, Wareham, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Care Access - Londonderry, Londonderry, New Hampshire
  - Care Access - North Conway, North Conway, New Hampshire
  - ActivMed Practices & Research, LLC., Portsmouth, New Hampshire
  - Internal Medicine Associates, Bridgeton, New Jersey
  - Clinilabs, Eatontown, New Jersey
  - Hunterdon Infectious Disease Specialists, Flemington, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Care Access - Hoboken, Hoboken, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Velocity Clinical Research, Binghamton, Binghamton, New York
  - Bassett Medical Center, Cooperstown, New York
  - Smith Allergy and Asthma Specialists, Cortland, New York
  - Care Access - Albany, Halfmoon, New York
  - Smith Allergy & Asthma Specialists, Horseheads, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - Velocity Clinical Research, Vestal, Vestal, New York
  - TruCare Internal Medicine & Infectious Disease, DuBois, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Central Erie Primary Care, Erie, Pennsylvania
  - Care Access - Mountaintop, Hazle Township, Pennsylvania
  - CCP - Kid's Way, Hermitage, Pennsylvania
  - Care Access - Kingston, Kingston, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Care Access - Pottsville, Pottsville, Pennsylvania
  - Care Access Mobile Site, Punxsutawney, Pennsylvania
  - Guthrie Medical Group, P.C., Sayre, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Care Access - Scranton, Scranton, Pennsylvania
  - Northeast Clinical Trials Group, Scranton, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Care Access - Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Care Access Mobile Site, Yeagertown, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Care Access Mobile Site, New Shoreham, Rhode Island
  - Care Access - Warwick, Warwick, Rhode Island
  - Care Access - Brattleboro - Putney Road, Brattleboro, Vermont
  - Care Access - Brattleboro, Brattleboro, Vermont
  - The University of Vermont Medical Center Inc., Burlington, Vermont
  - Care Access - Middlebury, Middlebury (village), Vermont
  - Amherst Family Practice, P.C., Winchester, Virginia
  - University of Wisconsin Carbone Cancer Center-University Hospital, Madison, Wisconsin
  - Marshfield Medical Center - Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (10):
  - Viable Clinical Research Corporation, Bridgewater, Nova Scotia
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Centricity Research Burlington Multispecialty, Burlington, Ontario
  - Milestone Research Inc., London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Stouffville Medical Research Institute Inc., Stouffville, Ontario
  - Centricity Research Toronto Manna Multispecialty, Toronto, Ontario
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
- Finland (9):
  - FVR, Tampereen rokotetutkimusklinikka, Tampere, Pirkanmaa
  - FVR, Turun rokotetutkimusklinikka, Turku, Southwest Finland
  - FVR, Etelä-Helsingin rokotetutkimusklinikka, Helsinki, Uusimaa
  - FVR, Itä-Helsingin rokotetutkimusklinikka, Helsinki, Uusimaa
  - FVR, Järvenpään rokotetutkimusklinikka, Jarvenpaa, Uusimaa
  - MeVac - Meilahti Vaccine Research Center, Helsinki
  - FVR, Kokkolan rokotetutkimusklinikka, Kokkola
  - FVR, Porin rokotetutkimusklinikka, Pori
  - Terveystalo Pulssi, Turku
- Germany (2):
  - AmBeNet GmbH, Leipzig, Saxony
  - Internistische Gemeinschaftspraxis Mainz, Mainz
- Amsterdam UMC, locatie AMC, Amsterdam, North Holland, Netherlands
- Poland (18):
  - Rodzinne Centrum Medyczne LUBMED, Luboń, Greater Poland Voivodeship
  - MICS Centrum Medyczne Torun, Torun, Kuyavian-Pomeranian Voivodeship
  - Przylądek Zdrowia, Krakow, Lesser Poland Voivodeship
  - Krakowski Szpital Specjalistyczny im. Jana Pawa II, Krakow, Lesser Poland Voivodeship
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska, Tarnów, Lesser Poland Voivodeship
  - Szpital im. Św. Jadwigi Śląskiej w Trzebnicy, Trzebnica, Lower Silesian Voivodeship
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Wroclaw, Lower Silesian Voivodeship
  - SZPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym, Łomianki, Masovian Voivodeship
  - Centrum Medyczne Lucyna Andrzej Dymek, Strzelce Opolskie, Opole Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Zespol Opieki Zdrowotnej w Boleslawcu, Bolesławiec
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Indywidualna Specjalistyczna Praktyka Lekarska Roman Spyra, Katowice
  - Centrum Badan Klinicznych Jagiellonskie Centrum Innowacji, Krakow
  - Krakowskie Centrum Medyczne, Krakow
  - NZOZ Praktyka Lekarza Rodzinnego Eskulap, Lublin
  - Przychodnia EuroMediCare Wroclaw Lowiecka, Wroclaw
  - Centrum Medyczne AD-MED Sp. z o. o. Przychodnia Dla Rodziny, Wroclaw
- Sweden (6):
  - Blekinge Tekniska Hogskola (BTH) (Blekinge Institute of Technology) - Karlskrona, Karlskrona, Blekinge LÄN [se-10]
  - CTC Karolinska, Solna, Stockholms LÄN [se-01]
  - Studieenheten Akademiskt Specialistcentrum, Stockholm, Stockholms LÄN [se-01]
  - CTC MTC, Uppsala, Uppsala LÄN [se-03]
  - ProbarE, Lund
  - Universitetssjukhuset Örebro, Örebro, Örebro LÄN [se-18]

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Dreyfus J, Munnangi S, Bengtsson C, Correia B, Figueiredo R, Stark JH, Zawora M, Riddle MS, Maguire JD, Jiang Q, Ianos C, Naredo Turrado J, Svanstrom H, Bailey S, DeKoven M. Background incidence rates of health outcomes in populations at risk for Lyme disease using US administrative claims data. Vaccine. 2024 Feb 15;42(5):1094-1107. doi: 10.1016/j.vaccine.2024.01.037. Epub 2024 Jan 22. PMID 38262807
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4601003